CLINICAL TRIAL: NCT02009774
Title: Accuracy of the Optical Diagnosis of Small Colonic Polyps Using the Nice Classification
Acronym: ADOPTION
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Dr. Peter Klare, MD, Technical University of Munich
Other Study IDs: ADOPTION
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-08

CONDITIONS: Colon Adenoma; Colorectal Carcinoma; Hyperplastic Polyp
Keywords: Colonoscopy; Adenoma detection rate; Narrow band imaging; Optical biopsy; Accuracy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controll group: Patients from the control group will be examined using a CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope. If colon polyps are detected optical diagnosis will be determined WITHOUT using the NBI function of the scope.
- Intervention: Patients from the control group will be examined using a CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope. If colon polyps are detected optical diagnosis will be determined WITH THE HELP OF the NBI function of the scope.
  Interventions: Procedure: NBI Function

INTERVENTIONS:
Procedure: NBI Function
  Other Names: NBI Function integrated in the CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope
  Groups: Intervention

SUMMARY:
Adenomas and hyperplastic polyps are polypoid lesion and may occur at any location in the colon. At the present moment, all polyps should be resected endoscopically, although only adenomas, but not hyperplastic polyps have the potential to develop colorectal cancer. This approach enables the conduction of microscopic investigations of the lesions. By today, only the pathological diagnosis can distinguish exactly between adenomas and hyperplastic polyps. Some studies have investigated the value of the socalled optical biopsy method. Optical biopsy means the visual assessment of the polyp and the determination of a diagnosis solely on behalf of optical criteria. This method is conducted in real time during colonoscopy. If it can be shown, that endoscopist using optical biopsy are able to predict histopathological diagnoses of colonic polyps sufficiently this would possibly lead to simplification of diagnostic procedures. For instance, it would be conceivable to resect hyperplastic polyps and small adenomas and discard them without further assessment by a pathologist. Gastroenterological societies demand for a 90 percent accordance between diagnoses set by endoscopists and pathologists as a prerequisite for the implementation of the optical biopsy method.

In this study we want to proof that the use of a new narrow-band imaging (NBI) tool (Exera III, Olmpus) is capable to rise accuracy of optically ascertained diagnoses of colonic polyps. NBI is a light filter tool which can be activated by pressing a button at the endoscope. NBI function leads to an endoscopic picture which appears blue and enables endoscopists to better assess surface structures and vascular patterns.

In a prospective randomised multicenter setting we plan to conduct colonoscopy in 380 patients. Half of the patients will be examined without use of NBI (control arm). In these cases colonoscopists will assess optical diagnosis of polyps without turning on the NBI tool. If polyps are detected in patients belonging to the intervention arm NBI will be used and optical diagnosis will be determined using the NICE (NBI International Colorectal Endoscopic) classification. All polyps will be resected and send to pathology for further microscopic assessment. After completing the trial we aim to compare accuracy of the optical diagnosis in both groups. Our hypothesis is, that by using the new NBI tool accuracy (accordance between optical and histopathological diagnosis) can be increased from 78% to 90%.

ELIGIBILITY:
Inclusion Criteria:

* medical indication for colonoscopy
* age >18 years
* written consent given by patient

Exclusion Criteria:

* age < 18 years
* patients denying written consent
* pregnant women
* ASA class IV, V and VI
* known contraindication for polyp resection
* indication for colonoscopy: preknown adenoma/polyp/carcinoma
* indication for colonoscopy: emergency (e.g. severe rectal bleeding)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the three participating study centers (Munich, Frankfurt, Berlin). Two of the three centers are tertiary referral-centres whereas the last one is a major regional hospital. All patients undergo colonoscopy for medical indications.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Accuracy optical biopsy | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)
  After obtaining the histopathological diagnosis of resected polyps (approximately 3 days - 2 weeks after colonoscopy ) accuracy of optical diagnosis can be determined

SECONDARY OUTCOMES:
Adenoma detection rate | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — Klinikum rechts der Isar der Technischen Universität München; Stefan von Delius, MD, Study Director — Klinikum rechts der Isar der Technischen Universität München; Jörg Albert, MD, Study Chair — Medizinische Klinik I University Hospital Frankfurt; Ellen C Nötzel, MD, Study Chair — Innere Medizin I, Sana Klinikum Lichtenberg
Locations (3):
- Germany (3):
  - II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria
  - Medizinische Klinik I des Universitätsklinikums Frankfurt, Frankfurt am Main, Hesse
  - Innere Medizin I am Sana Klinikum Lichtenberg, Berlin, State of Berlin

REFERENCES:
- [Derived] Klare P, Haller B, Wormbt S, Notzel E, Hartmann D, Albert J, Hausmann J, Einwachter H, Weber A, Abdelhafez M, Schmid RM, von Delius S. Narrow-band imaging vs. high definition white light for optical diagnosis of small colorectal polyps: a randomized multicenter trial. Endoscopy. 2016 Oct;48(10):909-15. doi: 10.1055/s-0042-110650. Epub 2016 Jul 22. PMID 27448051